CLINICAL TRIAL: NCT02422732
Title: Functional Magnetic Resonance Imaging and Reading Deficit in Children With NF1 Children
Brief Title: Functional Imaging and Reading Deficit in Children With NF1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 08 154 02; 2008-A01493-52 (Registry Identifier: ID-RCB)
Record Dates: First submitted 2015-03-27; First posted 2015-04-21 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Neurofibromatosis Type 1
Keywords: NF1; Children; Reading disability; Morphological and functional MRI; Genetic analysis
MeSH Terms: conditions — Neurofibromatosis 1; Dyslexia | interventions — Genetic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Children with reading disability (Other): Children with NF1, with reading disability if their performances on reading assessment (Alouette Test) present a delay of at least 18 months, will have Neuropsychological assessments, morphological and functional MRI (fMRI) and genetic analysis
  Interventions: Other: Neuropsychological assessments; Radiation: morphological and functional MRI (fMRI); Genetic: genetic analysis
- Children without reading disability (Other): Children with NF1, without reading disability if their performances on reading assessment (Alouette Test) present a less than 18-month delay, will have Neuropsychological assessments, morphological and functional MRI (fMRI) and genetic analysis.
  Interventions: Other: Neuropsychological assessments; Radiation: morphological and functional MRI (fMRI); Genetic: genetic analysis

INTERVENTIONS:
Other: Neuropsychological assessments — IQ (WISC-IV)
  Reading tests (reading accuracy, reading speed, reading comprehension and strategy):
  Alouette, Lobrot, Odedys tests. Visuo-spatial skill (JLO, Thurston, CORSI tests) Attention (CPT 2, CBCL) Receptive oral language (EVIP)
Radiation: morphological and functional MRI (fMRI) — The fMRI will consider on the acquisition of a 3D anatomical sequence in T1 high resolution in axial slices of 1mm with an acquisition time of 10 min and a T2 sequence and a "Flair" to allow UBO location.
Genetic: genetic analysis — Blood collection in 3 tubes (2 PAXgen® and 1 EDTA) and analysis to study the NF1 gene deletion.

SUMMARY:
A monocenter pilot study on the acceptability and feasibility of a functional MRI protocol in children with NF1 with or without reading disabilities.

DETAILED DESCRIPTION:
The principal aim of the study is to highlight the activation of brain area involved phonological and visuo-spatial processing in children with NF1 with or without reading disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age included between 8 and 12 years
* Child presenting a type 1 neurofibromatosis according to 2 criteria in the following criteria list :

  * At least 6 café au lait spots
  * 2 or more neurofibromas or 1 plexiform neurofibroma
  * axillary or inguinal freckling
  * 1 optic nerf glioma
  * 2 or more Lisch nodules
  * 1 osseous lesion as sphenoid dysplasia or thinning of the long bone cortex with or without pseudarthrosis
  * 1 A first degree relative (parent, sibling, or offspring) with NF1 by the above criteria
* Membership in a national insurance
* Consent of the child and the parents

Exclusion Criteria:

* Mental retardation (QI T < 70)
* Treated or untreated epilepsy
* Visual deficit (visual Acuteness < 4/10
* Presence of a symptomatic optic glioma
* Presence of a brain tumor.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2009-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Percentage of children performing in full the protocol functional MRI | day 1
  Study the acceptability and feasibility of a functional MRI protocol in children with NF1 with or without reading disabilities.

SECONDARY OUTCOMES:
blood flow in milliliters per minute | day 1
  Comparison of brain activations involved in phonological and visuo-spatial processing in 2 groups in children with NF1.
  1 group with reading disability and 1 group without reading disability Search for a link between the presence of a large deletion of the gene and learning disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Yves Chaix, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France